CLINICAL TRIAL: NCT03635931
Title: Efficiency of Concentrated Growth Factor in the Surgical Treatment of Multiple Adjacent Papillary Losses: a Controlled, Examiner-blinded Clinical Study
Brief Title: Surgical Treatment With Concentrated Growth Factor for Multiple Papillary Losses
Acronym: CGF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Collaborators: Ankara University (Other)
Responsible Party: Principal Investigator, Zeynep Turgut Çankaya, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 36290600
Record Dates: First submitted 2018-08-13; First posted 2018-08-17 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Papilla, Dentinal; Calcification
Keywords: CGF; lost interdental papilla
MeSH Terms: conditions — Calcinosis

STUDY DESIGN:
Intervention Model Description: The test and control group was formed of patients with adjacent papillary defects In test group, elective minimally invasive surgery for papillary regeneration with CGF was performed. A control group was formed of patients with adjacent papillary defects who were not included to have surgical treatment.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concentrated Growth Factor (Active Comparator): plaque control, scaling and root planing if required, surgical application of CGF
  Interventions: Procedure: Concentrated Growth Factor
- Control Group (No Intervention): plaque control, scaling and root planing if required

INTERVENTIONS:
Procedure: Concentrated Growth Factor — surgical treatment with CGF for papilla regeneration
  Arms: Concentrated Growth Factor

SUMMARY:
The aim of this study was to evaluate the efficacy of concentrated growth factor (CGF) in applied in the regenerative treatment of multiple adjacent papillary black triangles (MAPBT) occured as a result of soft tissue loss. Interdental papillary regeneration was evaluated with the change in the area of interproximal spaces calculated on each of the intraorally scanned images obtained with digital impressions of the interproximal space with irregular borders.This controlled, examiner-blinded, clinical study included of 40 patients with 120 open embrasures which resulted from papillary loss in adjacent teeth in the anterior maxillary esthetic zone resulting in black triangles (BTs). Then patients were randomly assigned to receive surgical regenerative periodontal treatment(test) or periodontal care(control)The test group was formed of 20 patients with 60 adjacent papillary defects . A control group was formed of 20 patients with 60 adjacent papillary defects.. A total of 480 images obtained with the digital impressions . Evaluations of the test group were made preoperatively and at 3, 6 and 12 months postoperatively. For the control group, oral hygiene instruction was provided. Control group is evaluated by the same procedure with test group but the surgical part is not performed. Lost interdental papillary area (PA)were calculated. In the test group, the percentage of papillary filling, the presence of keratinized gingiva, the thickness of papillary gingiva, blood thrombocyte count and mean platelet volume values(MPV) were recorded.

DETAILED DESCRIPTION:
The treatment of open gingival embrasures, which are also known as black triangles (BT) or black holes, and cause esthetic, functional and phonetic problems in the anterior region, has become an area of interest in current periodontal treatment.Surgical, non-surgical and prosthetic methods are applied in the treatment of BT, which can be seen in more than half of adults. This study aimed to evaluate the efficacy of concentrated growth factor (CGF) in regenerating interdental papillary of multiple adjacent papillary black triangles (MAPBT) occured as a result of soft tissue loss. Interdental papillary regeneration was evaluated with the change in the area of interproximal spaces calculated on each of the intraorally scanned images obtained with digital impressions of the interproximal space with irregular borders.

This controlled, examiner-blinded, randomized clinical study included 160 teeth of 40 patients with 120 open embrasures which resulted from papillary loss in adjacent teeth in the anterior maxillary esthetic zone resulting in black triangles (BTs). The test group was formed of 20 patients with 60 adjacent papillary defects undergoing minimally invasive surgery for papillary regeneration with CGF. A control group was formed of 20 patients with 60 adjacent papillary defects who were not included surgical treatment. A total of 480 images obtained with the digital impressions method of each interdental papillary region in each patient were uploaded to a special software. Evaluations of the test group were made preoperatively and at 3, 6 and 12 months postoperatively. For the control group, oral hygiene instruction was provided. Control group is evaluated by the same procedure with test group but the surgical part is not performed. Lost interdental papillary area (PA)were calculated between the two central teeth, between the lateral and central teeth, and between the lateral and canine teeth prior to the treatment and at pro-treatment periods of 3, 6 and 12 months in both of the groups. In the test group, the percentage of papillary filling, the presence of keratinized gingiva, the thickness of papillary gingiva, blood thrombocyte count and MPV values were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of interdental papillary losses in the maxillary anterior teeth, between the adjacent central teeth, the central and lateral teeth and the lateral and canine teeth
* The presence of a contact point in the maxillary anterior teeth
* optimal facial keratinized gingiva/ keratinized gingiva must be more than 2mm

Exclusion Criteria:

* pregnancy or
* breast-feeding,
* palatal and gingival recession,
* attachment loss,
* high labial frenulum.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-07-30 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-08-12 (Actual)

PRIMARY OUTCOMES:
change in the percentage of papillary fill(PF) | Change from 3 months percentage of papillary fill at 6 months
  The percentage of PF was also calculated as ([ Lost Papillary area(PA) preoperation - PA postoperation] / PA preoperation) x 100%.

CONTACTS AND LOCATIONS:
Overall Officials: zeynep Turgut Çankaya, PhD,Dr, Principal Investigator — Gazi University, Faculty of Dentistry,Department of Periodontology
Locations (1):
- Gazi University Faculty of Dentistry Department of Periodontology, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No